CLINICAL TRIAL: NCT00250380
Title: The Study on Profile and Genetic Factors of Aspirin Resistance (ProGEAR Study)-A Prospective Multicenter Cohort Study-
Brief Title: The Study on Profile and Genetic Factors of Aspirin Resistance (ProGEAR Study)
Status: Completed | Type: Observational
Sponsor: Ministry of Health, Labour and Welfare, Japan (Other Government)
Collaborators: The National Institute of Biomedical Innovation (Unknown)
Responsible Party: Principal Investigator, Toshiyuki Miyata, Director, National Cerebral and Cardiovascular Center, Japan
Other Study IDs: H17-CV(Seishu)-002
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Coronary Disease; Cerebral Infarction; Ischemic Attack, Transient
Keywords: Aspirin; Platelet Aggregation Inhibitors
MeSH Terms: conditions — Coronary Disease; Cerebral Infarction; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine the clinically meaningful definition and prevalence of aspirin resistance based on data linking aspirin-dependent laboratory tests to recurrent vascular events in cardiovascular patients taking aspirin.

DETAILED DESCRIPTION:
Primary Outcomes: The primary endpoint is the composite outcomes of cerebral infarction, transient ischemic attack, myocardial infarction, unstable angina, percutaneous coronary angiography, thromboembolism, and death caused by cardiovascular disease.

Secondary Outcomes: Platelet aggregation induced by collagen and arachidonic acid, serum thromboxane B2, urine 11-dehydrothromboxane B2, platelet thrombus formation under flow conditions (sub-study only at the National Cardiovascular Center)

The primary objective of this study is to determine the markers for aspirin resistance. To achieve this objective, platelet aggregation, serum thromboxane B2, and urine 11-dehydrothromboxane B2 are measured in patients receiving usual therapeutic doses of aspirin, who experienced acute coronary syndrome, cerebral infarction, or transient ischemic attack occurred in a period between the past 1 month and the past 2 years. This is a multi-center, prospective study.

ELIGIBILITY:
Inclusion Criteria:

Adult males or females who met the criteria listed below:

* Patients who had acute coronary syndrome, cerebral infarction (except cardioembolic stroke), or transient ischemic attack between past 28 days and the past 2 years
* patients who receive long-term aspirin therapy (at least 28 days)
* Patients who are >=20 years of age
* Patients willing and able to give written informed consent

Exclusion Criteria:

* Malignancy or suspected malignancy
* Patients who showed platelet counts less than 100,000/uL or more than 450,000/uL
* Congenital bleeding tendency
* Patients who receive other antiplatelet drugs or warfarin
* Patients with atrial fibrillation
* Patients who received surgical operation or catheter intervention within the past 2 weeks
* Patients who received anticoagulation drug therapy including heparin ( low-molecular weight heparin) and danaparoid.
* Patients with more than modified Rankin scale 4

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: out-patient clinic
Sampling Method: Probability Sample
Enrollment: 583 (Actual)
Dates: Start 2005-11; Primary Completion 2010-06 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toshiyuki Miyata, PhD, Principal Investigator — National Cardiovascular Center, Research Institute,; Shigeki Miyata, MD, Principal Investigator — National Cerebral and Cardiovascular Center, Japan; Kazuo Minematsu, MD, Principal Investigator — National Cerebral and Cardiovascular Center, Japan; Masafumi Kitakaze, MD, PhD, Principal Investigator — National Cerebral and Cardiovascular Center, Japan; Kazuyuki Nagatsuka, MD, PhD, Principal Investigator — National Cerebral and Cardiovascular Center, Japan; Atsushi Kawamura, MD, PhD, Principal Investigator — National Cerebral and Cardiovascular Center, Japan; Akiko Kada, MPH, Principal Investigator — National Cerebral and Cardiovascular Center, Japan; Shinichiro Uchiyama, MD, Principal Investigator — Tokyo Women's Medical University; Takehiko Nagao, MD, PhD, Principal Investigator — Tokyo Metropolitan Ebara Hospital; Naohisa Hosomi, MD, PhD, Principal Investigator — Kagawa University School of Medicine; Takemori Yamawaki, MD, PhD, Principal Investigator — Nagoya City University Graduate School of Medical Science; Kazumi Kimura, MD, PhD, Principal Investigator — Kawasaki Medical School; Kozue Saito, MD, Principal Investigator — Nara Medical University; Hiroshi Nakane, MD, Principal Investigator — National Fukuoka-Higashi Medical Center; Jyoji Nakagawara, MD, Principal Investigator — Nakamura Memorial Hospital; Shinya Goto, MD, Principal Investigator — Tokai University School of Medicine; Takaaki Isshiki, MD, Principal Investigator — Teikyo University; Kazuo Kitagawa, MD, Principal Investigator — Osaka University Graduate School of Medicine; Kazuomi Kario, MD, Principal Investigator — Jichi Medical School; Hideo Wada, MD, PhD, Principal Investigator — Mie University Graduate School of Medicine; Ken Nagata, MD, Principal Investigator — Research Institute for Brain and Blood Vessels Akita; Koichi Kaikita, MD, Principal Investigator — Kumamoto University Graduate School of Medicine; Keiji Tanaka, MD, Principal Investigator — Nippon Medical School Hospital; Akira Hattori, MD, Principal Investigator — Sado Hospital; Eisuke Furui, MD, PhD, Principal Investigator — Kohnan Hospital; Yoshihiko Saito, MD, PhD, Principal Investigator — Nara Medical University; Satoshi Ueno, MD, Principal Investigator — Nara Medical University; Yasuo Katayama, MD, Principal Investigator — Nippon Medical School Hospital; Takeo Abumiya, MD, Principal Investigator — Hokkaido Neurosurgical Memorial Hospital; Masakatsu Nishikawa, MD, Principal Investigator — Mie University Graduate School of Medicine; Shin Takiuchi, MD, PhD, Principal Investigator — Higashi Takarazuka Satoh Hospital; Hideyuki Ohnishi, MD, Principal Investigator — Ohnishi Neurological Center
Locations (23):
- Japan (23):
  - Research Institute for Brain and Blood Vessels Akita, Akita, Akita
  - National Fukuoka-Higashi Medical Center, Koga, Fukuoka
  - Hokkaido Neurosurgical Memorial Hospital, Sapporo, Hokkaido
  - Nakamura Memorial Hospital, Sapporo, Hokkaido
  - Ohnishi Neurological Center, Akashi, Hyōgo
  - Higashi Takarazuka Satoh Hospital, Takarazuka, Hyōgo
  - Kagawa University School of Medicine, Kida-gun, Kagawa-ken
  - Tokai University School of Medicine, Isehara, Kanagawa
  - Kumamoto University Graduate School of Medicine, Kumamoto, Kumamoto
  - Mie University Graduate School of Medicine, Tsu, Mie-ken
  - Kohnan Hospital, Sendai, Miyagi
  - Nagoya City University Graduate School of Medical Sciences, Nagoya, Nagoya
  - Nara Medical University, Kashihara, Nara
  - Sado Hospital, Sado, Niigata
  - Kawasaki Medical School, Kurashiki, Okayama-ken
  - Osaka University Graduate School of Medicine, Suita, Osaka
  - National Cardiovascular Center, Suita, Osaka
  - National Hospital Organization Ureshino Medical Center, Fujitsu-gun, Saga-ken
  - Jichi Medical School, Kawachi-gun, Tochigi
  - Nippon Medical School Hospital, Tokyo, Tokyo
  - Tokyo Metropolitan Ebara Hospital, Tokyo, Tokyo
  - Tokyo Women's Medical University, Tokyo, Tokyo
  - Teikyo University, Tokyo, Tokyo